CLINICAL TRIAL: NCT03913832
Title: Magic Touch Sirolimus Coated Balloon (Concept Medical) Versus SeQuent Pease Neo Paclitaxel Coated Balloon (Bbraun) for the Treatment of de Novo Coronary Artery Lesions in Small Vessels
Brief Title: TReAtmeNt of Small Coronary Vessels: MagicTouch Sirolimus Coated Balloon
Acronym: TRANSFORM I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Concept Medicals BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 180013
Record Dates: First submitted 2019-03-25; First posted 2019-04-12 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease; DCB
Keywords: small vessel; sirolimus; drug coating balloon
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sirolimus drug coated balloon (SCB) (Experimental): Magic TouchTM (Concept Medical) is a sirolimus drug coated balloon (SCB)
  Interventions: Device: sirolimus drug coated balloon (SCB)
- paclitaxel releasing coronary balloon catheter. (Active Comparator): SeQuent PleaseTM (B. Braun Melsungen AG, Vascular Systems,Berlin, Germany) is a paclitaxel releasing coronary balloon catheter
  Interventions: Device: paclitaxel releasing coronary balloon catheter

INTERVENTIONS:
Device: sirolimus drug coated balloon (SCB) — Magic TouchTM (Concept Medical) is a sirolimus drug coated balloon (SCB) for PCI, based on a polymer-free and Nano based drug delivery technology. Magic Touch SCB is a product of CMI proprietary drug delivery technology "Nanolute". It is indicated (CE approved) for ISR, small vessels, bifurcation lesions & de novo lesions.
  Arms: sirolimus drug coated balloon (SCB)
Device: paclitaxel releasing coronary balloon catheter — SeQuent PleaseTM (B. Braun Melsungen AG, Vascular Systems,Berlin, Germany) is a paclitaxel releasing coronary balloon catheter.
  Arms: paclitaxel releasing coronary balloon catheter.

SUMMARY:
The study is a prospective, multinational (Italy, Ireland and UK), multicenter, randomised Clinical Trial that compares the efficacy and performance of two drug coated balloon (DCB), the MAGIC TOUCH sirolimus coated balloon (Concept Medical) and SeQuent Please paclitaxel coated balloon (B Braun). The objective of the study is to compare angiographic outcomes of Magic TouchTM sirolimus coated balloon (Concept Medical) versus SeQuentTM paclitaxel coated balloon (Bbraun) for the treatment of de novo coronary artery lesions in small vessels (≤2.75 mm) with respect to Net Gain (mm) at 6 months follow-up

DETAILED DESCRIPTION:
A prospective, randomized, multi-centre study in subjects with small vessels, i.e. at least one de-novo lesion in a small vessel (≤2.75mm). Vessel size will be determined first by QCA on-line (screening, pre-procedure). If, based on QCA on-line the vessel size pre-procedure is ≤2.75mm and following a successful pre-dilatation (i.e. no angiographic dissections type CDEF and TIMI>2), the subject will be randomized in a 1:1 fashion to Magic Touch or SeQuent Please Neo. OCT will be performed post pre-dilatation (guidance) prior to drug coated balloon (DCB) treatment. The DCB balloon size will be selected based on OCT measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years
2. Patient with chronic stable angina or stabilized acute coronary syndromes with normal cardiac biomarker values

   Note: For patients showing elevated Troponin (e.g. non-STEMI patients) at baseline (within 72h pre-PCI) an additional blood sample must be collected prior to randomization to confirm that:
   * hs-cTn or Troponin I or T levels are stable, i.e. the value should be within 20% range of the value found in the first sample at baseline, or have dropped
   * CK-MB and CK levels are within normal range If hs-cTn or Troponin I or T levels are stable or have dropped, the CK-MB and CK levels are within normal ranges, and the ECG is normal, the patient may be included in the study.
3. The patient has a planned intervention in one or two separate major epicardial territories (LAD, LCX or RCA) and has at least one de-novo lesion in a small vessel (≤2.75mm by QCA prior to pre-dilatation)
4. Target lesion length ≤30 mm
5. Able to understand and provide informed consent and comply with all study procedures including 6 months angiographic follow-up
6. Patient must have completed the follow-up phase of any previous study

Exclusion Criteria:

1. Patient is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential)
2. Evidence of ongoing acute myocardial infarction (AMI) in ECG and/or elevated cardiac biomarkers (according to local standard hospital practice) have not returned within normal limits at the time of procedure
3. Known contraindication or hypersensitivity to sirolimus, paclitaxel, or to medications such as aspirin, heparin, and all of the following four medications: clopidogrel bisulfate, ticlopidine, prasugrel, ticagrelor
4. Patient suffered from stroke/TIA during the last 6 months
5. LVEF <30%
6. Platelet count <100,000 cells/mm3 or >400,000 cells/mm3, a WBC of <3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis)
7. Known renal insufficiency (e.g. serum creatinine >2.5mg/dL, or creatinine clearance ≤30 mL/min), or subject on dialysis, or acute kidney failure (as per physician judgment)
8. Patient undergoing planned surgery within 6 months with the necessity to stop DAPT
9. History of bleeding diathesis or coagulopathy
10. The patient is a recipient of a heart transplant
11. Concurrent medical condition with a life expectancy of less than 12 months
12. The patient is unwilling/not able to return for angiographic recatherisation at 6 month follow-up
13. Currently participating in another trial and not yet at its primary endpoint.

    Angiographic exclusion criteria:
14. The patient has a planned intervention in three separate major epicardial territories (3 vessel disease)
15. The patient has a planned intervention in the left-main plus two separate major epicardial territories (left-main plus 2 vessel disease)
16. Target vessel size >2.75 mm (by QCA)
17. Target vessel size <2.00 mm (by QCA)
18. Target lesion has a total occlusion or TIMI flow <2
19. Target lesion in left main stem
20. The target vessel contains visible thrombus
21. Aorto-ostial target lesion (within 3 mm of the aorta junction)
22. Moderate-severe tortuous, calcified or angulated coronary anatomy of the target vessel that in the opinion of the investigator would result in suboptimal imaging or excessive risk of complication from placement of an OCT catheter
23. Lesion is located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2023-03-10 (Estimated); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
Net Gain (mm) In-segment | 6 Months
  The primary endpoint is in-segment (balloon treated area) Net Gain (mm) at 6 months post-procedure.

SECONDARY OUTCOMES:
Device success | Post procedure (Right after the treatment with drug coated balloon)
  Successful delivery and inflation within 45 seconds of the allocated DCB device at the intended target lesion during an attempt with a DCB not previously used (first use) and successful withdrawal of the device system with attainment of final in-lesion residual stenosis of <30% (by Quantitative Coronary angiography).
Procedure Success | Post procedure (Right after the treatment with drug coated balloon)
  Successful delivery and inflation within 45 seconds of the allocated DCB device at all intended target lesion(s) during an attempt with a DCB not previously used (first use) and successful withdrawal of the device system with attainment of final in-lesion residual stenosis of <30% (by QCA) without the occurrence of TLF during the index procedure hospital stay).
Acute/subacute/early/late vessel closure/thrombosis | 1, 6 months and 12 Months
  Closure by restenosis or thrombosis (diameter stenosis of 100% and/or TIMI grade 0).
Angiographic outcomes: late lumen loss | 6 months
  The difference between the minimum lumen diameter (MLD) immediately after index procedure and the MLD at follow-up as measured in (preferable) identical orthogonal views (MLDpost - MLDfup).
Angiographic outcomes:Minimal lumen diameter | 6 months
  The smallest lumen diameter in the segment of interest
Angiographic outcomes: Percent diameter stenosis | 6 months
  The percentage of luminal narrowing of vessel segment of interest
Angiographic outcomes: Restenosis rate | 6 months
  Restenosis is defined as ≥50% diameter stenosis at follow-up.
Device oriented Composite Endpoint (DoCE / TLF): Cardiac death | 1, 6 months and 12 Months
  Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all study procedure related deaths including those related to concomitant treatment.
Device oriented Composite Endpoint (DoCE / TLF): Target vessel: myocardial infarction (TV-MI) | 1, 6 months and 12 Months
  The term myocardial injury should be used when there is evidence of elevated cardiac troponin values (cTn) with at least one value above the 99th percentile upper reference limit (URL) TV-MI: Myocardial Infarction not clearly attributable to a non-target vessel.
Device oriented Composite Endpoint (DoCE / TLF): clinically indicated target lesion revascularization(TLR) | 1, 6 months and 12 Months
  TLR is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Serruys, Dr, Study Chair — NUIG Imaging CoreLab; Bernardo Cortese, Dr, Study Chair — Fondazione RIC
Locations (6):
- Galway University Hospital, Galway, Ireland
- Italy (4):
  - Maria Cecilia Hospital spa, Cotignola, Emilia-Romagna
  - I.R.C.C.S. Policlinico San Donato, San Donato Milanese, Lombardy
  - AOUC Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany
  - Istituto Clinico Humanitas, Rozzano
- Heart of England NHS Trust, Heartlands Hospital, Birmingham, United Kingdom

REFERENCES:
- [Derived] Ono M, Kawashima H, Hara H, Katagiri Y, Takahashi K, Kogame N, Wykrzykowska JJ, Piek JJ, Doshi M, Sharif F, Onuma Y, Colombo A, Serruys PW, Cortese B. A Prospective Multicenter Randomized Trial to Assess the Effectiveness of the MagicTouch Sirolimus-Coated Balloon in Small Vessels: Rationale and Design of the TRANSFORM I Trial. Cardiovasc Revasc Med. 2021 Apr;25:29-35. doi: 10.1016/j.carrev.2020.10.004. Epub 2020 Oct 17. PMID 33109476
- See also: Study website — http://transform1trial.com/